CLINICAL TRIAL: NCT04739527
Title: An Open Label, Phase 1 Study to Evaluate the Safety, Feasibility and Immunogenicity of an Allogeneic, Cell-based Vaccine (DCP-001) in High Grade Serous Ovarian Cancer Patients After Primary Treatment
Brief Title: Phase 1 Study to Evaluate the Safety, Feasibility and Immunogenicity of an Allogeneic, Cell-based Vaccine (DCP-001) in High Grade Serous Ovarian Cancer Patients After Primary Treatment
Acronym: ALISON
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Mendus (Industry)
Responsible Party: Principal Investigator, Hans W. Nijman, MD PHD, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALISON-UMCG-01
Record Dates: First submitted 2021-01-08; First posted 2021-02-04 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label phase I study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients receiving 4 bi-weekly vaccinations with 25E6 cells/vaccination of DCP-001, and 2 booster vaccinations with 10E6 cells/vaccination
  Interventions: Biological: DCP-001

INTERVENTIONS:
Biological: DCP-001 — allogeneic dendritic cell vaccine

SUMMARY:
Phase I study to evaluate safety and systemic immunogenicity of the DCP-001 vaccine in patients with high grade serous ovarian cancer after primary treatment.

DETAILED DESCRIPTION:
This is a first phase I study in HGSOC patients with primary disease eligible for standard of care treatment with either; complete or optimal primary cytoreductive surgery followed by 6 cycles of adjuvant chemotherapy (carboplatin/paclitaxel); or 3 cycles of neoadjuvant chemotherapy (carboplatin/paclitaxel) followed by complete or optimal cytoreductive interval surgery and 3 additional cycles carboplatin/paclitaxel.

In the current study, DCP-001 vaccinations will be scheduled after standard of care treatment, starting 6 weeks after the last cycle of chemotherapy.

Patients will receive 4 vaccinations containing 25E6 DCP-001 cells per vaccination followed by 2 additional booster vaccinations of 10E6 cells. Each patient will be followed up for 24 months. Safety will be monitored throughout the study. Systemic immune responses are determined by standard immune assays using peripheral blood mononuclear cells (PBMCs) and serum collected before, during and after vaccinations. Progression of disease will be monitored according to standard-of-care follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Primary HGSOC patients (FIGO stage 3B to IV) who completed primary treatment defined as:

  * primary debulking surgery (complete / optimal) and 6 cycles of adjuvant chemotherapy (carboplatin/paclitaxel)
  * 3 cycles of neo-adjuvant chemotherapy (more NACT cycles to improve surgical outcome are allowed) followed by interval debulking surgery (complete / optimal) and 3 cycles of adjuvant chemotherapy (carboplatin/paclitaxel)
* Serum level CA125 < 35 U/mL
* Age ≥ 18 years
* Signed informed consent form (ICF) in accordance with institutional and regulatory guidelines

Exclusion Criteria:

* History of a second malignancy except for curatively treated low-stage tumors with a histology that can be differentiated from the epithelial OC type
* Patients must have no ongoing or recent evidence (within the last 5 years) of significant autoimmune disease that required treatment with systemic immunosuppressive treatments which may suggest risk for immune-related adverse events (irAEs).

Note: Patients with autoimmune-related hyperthyroidism, autoimmune-related hypothyroidism who are in remission, or on a stable dose of thyroid-replacement hormone, vitiligo, or psoriasis may be included.

* Patients must have no uncontrolled infection with human immunodeficiency virus, hepatitis B or hepatitis C infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection. Mild cancer-related immunodeficiency (such as immunodeficiency treated with gamma globulin and without chronic or recurrent infection) is allowed.

  * Patients with known HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
  * Patients with known hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving antiviral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of trial treatment.
  * Patients who are known hepatitis C virus antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
* Liver or renal function abnormalities that are considered to be clinically relevant by the investigator.
* Abnormal blood levels (neutropenia among other things) due to chemotherapy that are considered to be clinically relevant by the investigator.

  * If so, blood levels will be repeated in 1-2 weeks, in case blood levels are normalized the patient is allowed to be included in the study. In case of persistent abnormal blood levels the patient will be excluded.
* Use of systemic continuous corticosteroid therapy (e.g. prednisone i.v. or p.o. >7.5 mg / day).
* Participation in a trial with another investigational drug within 30 days prior to the enrolment in this trial
* Any condition that in the opinion of the investigator could interfere with the conduct of the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline DCP_001 vaccine antigen-specific T cells in the peripheral blood (systemic induction / expansion of DCP_001 vaccine antigen-specific T cells) | A PBMC collection is planned at baseline, before start treatment. Further PBMC collections are scheduled during (4 times) and after the vaccinations.
  Systemic DCP-001 vaccine specific response is measured by the number of patients with de novo or increased immune responses based on IFNƴ ELISpot assay in any or more of the post-vaccination PBMC samples to at least one of the following DCP-001 vaccine antigens compared to baseline: WT-1, Survivin, RHAMM or PRAME, specific cancer testis antigens as NY-ESO1 and MAGE3.

SECONDARY OUTCOMES:
Safety and tolerability of the repetitive doses of the DCP-001 vaccine | Up to 28 days after last vaccination
  Number of patients with AEs, and SAEs
Recurrence free survival (RFS) | Up to 2 years from disease diagnosis
  RFS defined as the number of patients alive without any progress or recurrence (local or regional, or distant) and death due to any cause
Overall survival (OS) | Up to 2 years from disease diagnosis
  OS defined as the number of patients alive, measured in months, up to 2 years from disease diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Hans W Nijman, MD/PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No